CLINICAL TRIAL: NCT01535820
Title: A Bioequivalence Study to Evaluate the Effect of an Adhesive Overlay on the Delivery of Contraceptive Hormones From ORTHO EVRA® in Healthy Women
Brief Title: The Effect of an Adhesive Overlay on the Delivery of Contraceptive Hormones From ORTHO EVRA® in Healthy Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100412; NRGEEPCON1017 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2012-02-15; First posted 2012-02-20 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; ORTHO EVRA; Contraceptive hormones; Transdermal patch; Progestin norelgestromin (NGMN); Estrogen ethinyl estradiol (EE); JNJ-93964; JNJ-622206

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment sequence AB (Experimental)
  Interventions: Drug: Treatment A: ORTHO EVRA patch (NGMN + EE) with an adhesive overlay; Drug: Treatment B: ORTHO EVRA patch (NGMN + EE) without an overlay
- Treatment sequence BA (Experimental)
  Interventions: Drug: Treatment A: ORTHO EVRA patch (NGMN + EE) with an adhesive overlay; Drug: Treatment B: ORTHO EVRA patch (NGMN + EE) without an overlay

INTERVENTIONS:
Drug: Treatment A: ORTHO EVRA patch (NGMN + EE) with an adhesive overlay — NGMN: type= exact number, unit= mg, number= 6, form= transdermal patch, route= transdermal use. EE: type= exact number, unit= mg, number= 0.75, form= transdermal patch, route= transdermal use. A single patch is applied to the buttock with an adhesive overlay applied over the transdermal contraceptive system for 7 days.
Drug: Treatment B: ORTHO EVRA patch (NGMN + EE) without an overlay — NGMN: type= exact number, unit= mg, number= 6, form= transdermal patch, route= transdermal use. EE: type= exact number, unit= mg, number= 0.75, form= transdermal patch, route= transdermal use. A single patch is applied to the buttock without an overlay for 7 days.

SUMMARY:
The purpose of this study is to assess the bioequivalence of the contraceptive hormones of ORTHO EVRA when the patch is applied with and without an adhesive overlay.

DETAILED DESCRIPTION:
This is a randomized (the study drug is assigned by chance), open-label (all people know the identity of the intervention), single-center, single-application, 2-way crossover study (participants receive different interventions sequentially during the trial) of ORTHO EVRA with and without an adhesive overlay. ORTHO EVRA is a combination transdermal (through the skin) contraceptive patch containing 6.00 mg of the progestin norelgestromin (NGMN) and 0.75 mg of the estrogen, ethinyl estradiol (EE). The participants will be randomly assigned to 1 of 2 possible treatment sequences to ensure that they receive both of the following treatments, 1 in each period: - Treatment A: ORTHO EVRA patch applied to the buttock with an adhesive overlay applied over the transdermal contraceptive system; - Treatment B: ORTHO EVRA patch applied to the buttock without an overlay. The study consists of a screening phase; an open-label treatment phase consisting of 2 single-application 7-day treatment periods; and end-of-study or withdrawal assessments done upon completion of the 240-hour pharmacokinetic sampling on Day 11 of Period 2 or upon withdrawal. Pharmacokinetic evaluations explore how the drug is absorbed in the body, distributed within the body, and how it is removed from the body over time. The two treatment periods will be separated by a washout period (period when receiving no treatment) of 21 days. During the study, safety and tolerability will also be assessed. The total duration of participation in the study for an individual will be approximately 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Body mass index (BMI) between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg and not more than 90 kg
* Must be surgically sterile with intact ovaries, abstinent, or, if sexually active, be practicing an effective method of non-hormonal birth control (eg, non-hormonal intrauterine device, double-barrier method, male partner sterilization) before entry and throughout the study
* Completed her last term pregnancy at least 90 days before admission to the study site
* History of regular menstrual cycles (occurring every 25 to 35 days)
* Must not be pregnant or lactating
* Blood pressure between 90 and 140 mmHg systolic (inclusive), and no higher than 90 mmHg diastolic
* Hemoglobin equal or more than 12.0 at screening

Exclusion Criteria:

* History of smoking or use of nicotine-containing substances
* Used steroid hormonal therapy within 30 days before admission to the study
* Received a Depo Provera® injection in the 6 months before admission to the study
* History or presence of disorders commonly accepted as contraindications to sex hormonal therapy
* History of or current clinically significant medical illness or any other condition that the investigator considers should exclude the patient or that could interfere with the interpretation of the study results

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
NGMN plasma concentrations (Periods 1 and 2) | At 0, 24, 48, 72, 120, 168, 171, 174, 180, 192, 204, 216, and 240 hours.
EE plasma concentrations (Periods 1 and 2) | At 0, 24, 48, 72, 120, 168, 171, 174, 180, 192, 204, 216, and 240 hours.

SECONDARY OUTCOMES:
Pharmacokinetic parameters of NGMN (Periods 1 and 2) | At 0, 24, 48, 72, 120, 168, 171, 174, 180, 192, 204, 216, and 240 hours.
  Pharmacokinetic parameters of NGMN as measured by AUC, Cmax, tmax, and Css.
Pharmacokinetic parameters of EE (Periods 1 and 2) | At 0, 24, 48, 72, 120, 168, 171, 174, 180, 192, 204, 216, and 240 hours.
  Pharmacokinetic parameters of EE as measured by AUC, Cmax, tmax, and Css.
Incidence of adverse events as a measure of safety and tolerability | Approximately 2 months
The number of patients with changes in clinical laboratory test values, physical examination results, and vital signs measurements | Approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Neptune City, New Jersey, United States